CLINICAL TRIAL: NCT06344858
Title: Characterization of the Temporal Profile of the Anti- Nociceptive Effect of an Intravenous Ketamine Bolus Using the Nociception Analgesia Index (ANI)
Brief Title: Characterization of the Temporal Profile of the Anti-nociceptive Effect of Ketamine Bolus Measured With ANI
Acronym: Keta-ANI
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 124/2021
Record Dates: First submitted 2024-02-05; First posted 2024-04-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Analgesia; Ketamine; Pharmacokinetic
Keywords: Ketamine; Analgesia; Target controlled infusion
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ketamine: In the preoperative room a vein of the forearm with preriferic access #18 will be established for the administration of general intravenous anesthesia and intraoperative fluids.
  In the operating room, after routine monitoring (Heart Rate, Non-Invasive Blood Pressure, Oxygen Saturometry), the sensor of the Nociception Analgesia Index (ANI) monitor will be installed from the right chest to the left 5th intercostal space.
  Wait XX time for calibration and capture of the electrocardiographic signal. The ANI value shall initially be measured and shall be considered as the reference value.
  Inject 0.1 mg/kg of ketamine (1 mg/ml) once, then inject 5 ml of physiological saline at the same rate.
  The time from ketamine administration until the ANI index rose above 50 (minimum appropriate nociception value) shall be recorded every 6 seconds.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — One bolus of ketammine
  Other Names: Analgesia using ketamine

SUMMARY:
Ketamine, an intravenous anesthetic, and analgesic agent has experienced a resurgence in its clinical application, particularly in subanesthetic doses. The aim of this observational study is to characterize the changes in the Nociception Analgesia Index (ANI) associated with the administration of an intravenous ketamine bolus using a Pharmacokinetic-Pharmacodynamic (PKPD) modeling approach. The pharmacokinetic parameters of the Domino model will be used to predict ketamine plasma concentrations after the bolus dose. An Emax model and a link model assuming a first order rate constant (ke0) will be used to fit the data. Modeling analysis will use the program NONMEM. It is expected to recruit a total of 20 patients between 40 and 80 years, ASA I, II or III, programmed for elective surgery with general anesthesia. ANI values will be recorded every 6 seconds for 5 minutes from the bolus dose.

DETAILED DESCRIPTION:
Ketamine was introduced into clinical practice in 1965 and has been widely used as an intravenous anesthetic and analgesic. In recent years there has been a resurgence in its use mainly using low intravenous doses as a multimodal analgesia strategy and attenuation of postoperative hyperalgesia. Its use in low doses as an analgesic has also grown in other areas such as in emergency medicine and in patients with chronic pain and neuropathic pain. While optimal analgesic doses are not well defined in general the recommended regimens range from 0.15 to 0.3 mg/kg bolus and infusions from 0.1 to 0.3 mg/kg/h.

Target-controlled infusion (TCI) is an intravenous anesthesia delivery technique that incorporates pharmacokinetic models in pump infusion algorithms to allow obtaining objective-stable concentrations of the drug in the plasma or effect site. The TCI mode effect site presents advantages over plasma-to-plasma TCI since plasma concentrations do not have a good correlation with the drug's effect in nonequilibrium scenarios. This modality is based on that TCI systems can be instructed to exceed the desired plasma concentration to accelerate the rate at which the drug's effect is achieved. For the pharmacokinetic model to perform this the parameter set has to have the ke0 which is the equilibrium constant between the plasma and the effect site. This parameter provides the necessary information of the time profile of the drug's effect to the model. These models are known as on-site effect models or PKPD models. The potential benefit of TCI to site effect is the most accurate titration of the desired effect. Moreover, these models allow us to better understand the temporal profile of the drug effect.

TCI has been used for ketamine administration in various settings, including critical care. The operating room, and studies in neuroscience. In routine practice, ketamine TCI is performed using the model described by Domino with plasma target concentrations lower than 1.2 ng/ml to obtain its anti-nociceptive effect. Currently ketamine TCI can only be used in plasma mode since ke0 for its analgesic effect has not been determined.

The analgesic monitor PhysioDolorisTM (MDoloris Medical Systems SAS, Lille, France) was developed to quantitatively evaluate the effects of nociceptive stimuli on analgesic/nociceptive balance (the balance between the sympathetic/parasympathetic nervous system) in the anesthetized patient. ANI monitoring provides information on physiological coding and processing of nociceptive stimuli by analyzing the high-frequency component of heart rate variation in relation to respiratory rate. During anesthesia, the nociception index values reflect whether analgesia is adequate and whether analgesia allows the maintenance of nociception-antinociception balance, in which parasympathetic activity predominates over sympathetic. This monitoring provides a promising and objective evaluation of nociception.

The aim of this observational study was to describe changes in the ANI value associated with the administration of an intravenous ketamine bolus in a group of patients scheduled for elective surgery under general anesthesia.

The hypothesis is that the anti-nociceptive effect of the drug can be characterized by changes in ANI associated with the administration of a ketamine bolus. Effect-site TCI will be possible by incorporating this information into the available ketamine pharmacokinetic models.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery with general anaesthesia
* Without premedication
* ASA I, II or III

Exclusion Criteria:

* Body weight greater than 120% of ideal weight
* Ingestion of sedatives of short or long action in the 48 hours before surgery
* People with a history of adverse effects to the drug under study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery with general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
To measure ANI values after ketamine bolus dose administration. | Every 6 seconds for 5 minutes after ketamine bolus
  The observed effect of ketamine is measured with the ANI monitor index in each patient (outcome is ANI values [ANI Units])
To determine the time maximum predicted concentrations in each patient | Every 6 seconds for 5 minutes after ketamine bolus
  The time from the start of ketamine administration until the maximum predicted ketamine plasma concentrations value will be determined in each patient (mg/L).
To determine the time to maximum effect of a bolus dose of ketamine | Every 6 seconds for 5 minutes after ketamine bolus
  The time from the start of ketamine administration until the maximum ANI index value will be determined in each patient (ANI Values/minutes)
To predict ketamine plasma concentrations values after ketamine bolus | Every 6 seconds for 5 minutes after ketamine bolus
  The expected maximum plasma concentrations mg/L. Wil be estimated using the pharmacokinetic parameters of Domino knowing the administered dose (0.1 mg/Kg).
To calculate the difference between the time of maximum ANI effect | At the minute of maximum effect
  With the time (minutes) maximum predicted concentrations and the ketamine plasma concentrations (mg/mL)

SECONDARY OUTCOMES:
Patient weight | Once before the procedure
  The patient's weight will be measured prior to the administration of the ketamine bolus, which will be described in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortinez, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided